CLINICAL TRIAL: NCT04637152
Title: Anti-Hypertensive Effect of Sacubitril/Valsartan in Resistant Hypertension: Randomized Clinical Trial - The HEVA Study
Brief Title: Sacubitril/Valsartan in Resistant Hypertension
Acronym: HEVA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital Geral Roberto Santos (Other)
Collaborators: Hospital Universitário Professor Edgard Santos (Other)
Responsible Party: Principal Investigator, Andre Rodrigues Duraes, Medical Director, Hospital Geral Roberto Santos
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HGeralRobertoSantos
Record Dates: First submitted 2020-11-14; First posted 2020-11-19 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Resistant Hypertension; Blood Pressure
Keywords: Resistant Hypertension; LCZ696; Blood pressure control; sacubitril/valsartan
MeSH Terms: interventions — sacubitril and valsartan sodium hydrate drug combination

STUDY DESIGN:
Intervention Model Description: It was adopted an equal allocation of patients to each treatment (i.e., 1:1 randomization)
Who Masked: Investigator
Masking Description: Single (Investigator)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A: Usual recommended therapy (No Intervention): Antihypertensive regimen based on the usual recommended (optimized) therapy.
- Group B: Sacubitril/Valsartan (Experimental): Suspension of ACE inhibitors - for at least 36h of the last dose - or ARB. Initial dosage: Sacubitril/valsartan 49mg/51mg, 1 tablet twice daily. Target dose (after two weeks): 97mg/103 mg, 1 tablet twice daily.
  Interventions: Drug: Sacubitril-Valsartan

INTERVENTIONS:
Drug: Sacubitril-Valsartan — Use of sacubitril/valsartan after suspension of ACE inhibitors or ARBs.
  Arms: Group B: Sacubitril/Valsartan

SUMMARY:
The present study aims to evaluate the antihypertensive effect of sacubitril/valsartan in patients with resistant hypertension compared to the use of recommended and optimized antihypertensive therapy, through a randomized clinical trial, over 12 weeks.

DETAILED DESCRIPTION:
Worldwide, millions of people are affected by the arterial hypertension system (SAH), so that the presence of resistant hypertension (RH) significantly influences a high cardiovascular morbidity and mortality compared to those with controlled SAH, thus corroborating the need for the development of agents antihypertensive drugs with favorable efficacy and safety profiles. It is known that they are currently using the combined therapy recommended for this group of patients, among them, a significant portion of individuals with RH are unable to achieve the goal of BP control (>140/90 mmHg) even though in regular use, being subject to the greatest risk of cardiovascular outcomes and morbidity and mortality. Approved by the FDA for use in heart failure with reduced ejection fraction with beneficial effects on morbidity and mortality, identified in previous studies, the sacubitril/valsartan molecule (LCZ696) or Entresto® is a molecular complex composed of the sacubitril prodrug activated after ingestion in sacubitrilate - neprilysin inhibitor - associated with valsartan, an angiotensin II type-1 (AT1) receptor antagonist, with vasodilating action, capable of reducing BP, sympathetic tone, with antifibrotic and anti-hypertrophic effects, in addition to natriuresis and diuresis. Considering the knowledge gap to the benefits to LCZ696 in the control of blood pressure in resistant hypertension, the objective of the present study is to evaluate the efficacy (reduction of ambulatory systolic and diastolic blood pressure) and safety (adverse events, hospitalization and cardiovascular death) of the use of sacubitril/valsartan in comparison to the antihypertensive therapy recommended and optimized by the current guidelines, in patients diagnosed with RH, over12 weeks, through a randomized clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Men or women, over 18;
* Diagnosed with resistant hypertension (using three or more antihypertensive agents of different classes - eg. angiotensin-converting enzyme inhibitor, angiotensin II receptor blocker, calcium channel blockers, loop and thiazide diuretics or potassium-sparing diuretics), at least 4 weeks before recruitment, with a BP that remains above the goal of 140/90 mmHg.

Exclusion Criteria:

* Secondary and treatable hypertension;
* History of angioedema; significant cerebrovascular disease;
* Active liver disease (alanine aminotransferase or aspartate aminotransferase > 2 times the upper limit of the normal range and)
* Kidney dialysis or kidney transplantation or serum creatinine> 1.5 times the upper limit of the normal range or CrCl <30 mL/min;
* Previous or current diagnosis of heart failure;
* Malignancy;
* Any significant laboratory abnormalities such as serum potassium > 5.5 mmol/L.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-11-11 (Actual); Primary Completion 2022-07-22 (Actual); Study Completion 2022-08-17 (Actual)

PRIMARY OUTCOMES:
achieving the blood pressure target of <140/90mmg and the reducing of the mean sitting systolic blood pressure (msSBP), mean sitting diastolic blood pressure (msDBP), and mean sitting pulse pressure (msPP) over an 8-week period. | 8 weeks
  2 co-primary outcomes
Secondary efficacy outcomes included BP reduction stratified by Sac-Val dose compared to standard therapy. | 8 weeks
  Secondary outcome

SECONDARY OUTCOMES:
Secondary safety outcomes included incidence of acute myocardial infarction, hospitalization, stroke, hypotension, angioedema, electrolyte disturbances, CKD progression, and CV mortality | 8 weeks
  Safety outcomes

CONTACTS AND LOCATIONS:
Locations (2):
- Brazil (2):
  - General Hospital Roberto Santos, Salvador, Estado de Bahia
  - Hospital Universitário Professor Edgard Santos, Salvador, Estado de Bahia

IPD SHARING:
Plan to Share IPD: Undecided